CLINICAL TRIAL: NCT03021642
Title: A Phase I, Open-label, Randomized, Cross-over Trial to Investigate the Relative Bioavailability of Two Tepotinib Film-Coated Tablet Formulations in Healthy Volunteers
Brief Title: Relative Bioavailability of Two Tepotinib Film-Coated Tablet Formulations in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: MS200095-0012; 2015-004369-95 (EudraCT Number)
Record Dates: First submitted 2017-01-12; First posted 2017-01-16 (Estimated); Results first posted 2019-01-25 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Healthy
Keywords: Healthy volunteer; Tepotinib; Mesenchymal-epithelial transition factor; Translocated promoter region

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- First Tepotinib Test, Then Tepotinib Reference (Experimental)
  Interventions: Drug: Tepotinib test (Treatment Period 1); Drug: Tepotinib reference (Treatment Period 2)
- First Tepotinib Reference, Then Tepotinib Test (Experimental)
  Interventions: Drug: Tepotinib reference (Treatment Period 1); Drug: Tepotinib test (Treatment Period 2)

INTERVENTIONS:
Drug: Tepotinib test (Treatment Period 1) — Subjects will be administered a single oral dose of test treatment of film-coated tepotinib tablet (1 * 500 mg tablet) in Treatment period 1 (Day 1)
  Arms: First Tepotinib Test, Then Tepotinib Reference
Drug: Tepotinib reference (Treatment Period 2) — Followed by a 21-day washout after Treatment period 1 (Day 1), subjects will be administered a single oral dose of reference treatment of film-coated tepotinib tablet (5 * 100 mg tablet) in Treatment period 2 (Day 22)
  Arms: First Tepotinib Test, Then Tepotinib Reference
Drug: Tepotinib reference (Treatment Period 1) — Subjects will be administered a single oral dose of reference treatment of film-coated tepotinib tablet (5 * 100 mg tablet) in Treatment period 1 (Day 1)
  Arms: First Tepotinib Reference, Then Tepotinib Test
Drug: Tepotinib test (Treatment Period 2) — Followed by a 21-day washout after Treatment period 1 (Day 1), subjects will be administered a single oral dose of test treatment of film-coated tepotinib tablet (1 * 500 mg tablet) in Treatment period 2 (Day 22)
  Arms: First Tepotinib Reference, Then Tepotinib Test

SUMMARY:
This is a Phase I, open label, randomized, crossover trial to investigate the relative bioavailability of tepotinib in healthy volunteers. Twenty-four volunteers will be randomized to one of the two treatment sequences: Sequence A: test, reference, Sequence B: reference, test. The reference treatment refers to the current Phase II film-coated tablet (5 * 100 milligram (mg) tepotinib film-coated tablets) and the test treatment to the new Phase III film-coated tablet (1 * 500 mg film-coated tepotinib tablet).

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and non-fertile, healthy female volunteers, 18 to 60 years of age (both inclusive) at the time of informed consent.
* Written informed consent given before any trial related activities are performed.
* Body weight greater than 50 kg and a body mass index (BMI) above 18 kilogram per meter square (kg/m^2) and below 30 kg/m^2 (BMI = weight [kg]/height [m^2]) at screening.
* Has vital signs in the following normal range:

  * Oral body temperature: 35.5 to 37.5 degree celsius (°C)
  * Blood pressure (BP) and pulse rate after at least 5 minutes of rest, measured in the supine position: Systolic blood pressure: 90 to 150 millimeter of mercury (mm Hg); Diastolic blood pressure: 40 to 90 mm Hg
  * Pulse rate: 35 to 110 beats per minute (bpm)
* Non-smoker (= 0 cigarettes, pipes, cigars, e-cigarettes, or others) for at least 6 months prior to screening
* Women must be postmenopausal for at least 2 years, as confirmed by luteinizing hormone (LH) and follicle-stimulating hormone (FSH) assessments performed at screening, or surgically sterile (that is, hysterectomy, oophorectomy). Pregnancy assessments will also be performed on female volunteers at screening and at admission.
* Males must agree to use and to have their female partners use highly effective medically acceptable methods of contraception during the period of participation in the trial and for at least 3 months after the last treatment administration. Men must refrain from donating sperm up to 3 months after the last treatment administration.
* Ability to understand the full nature and purpose of the trial, including possible risks and adverse effects; ability to cooperate with the Investigator and to comply with the requirements of the entire trial, including dietary restrictions.

Exclusion Criteria:

* Any condition, including findings in the medical history, physical examination or in pretrial assessments that in the opinion of the Investigator, constitutes a risk or a contraindication for the participation of the volunteer in the trial or that could interfere with the trial objectives, conduct or evaluation.
* Any clinically relevant abnormality in the results of the screening safety laboratory parameters. Specifically Alanine transaminase (ALT), aspartate aminotransferase (AST), total bilirubin, Alkaline phosphatase (ALP), amylase, and lipase must not exceed the upper limit of the normal range.
* Any clinically relevant abnormality on the 12-lead electrocardiogram recording.
* Positive result from virology tests for hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (anti-HCV), or human immunodeficiency virus antibody (anti-HIV 1 and 2) at screening.
* History of clinically relevant renal, cardiovascular, and pulmonary disease, or endocrinology disorder.
* History of clinically relevant gastrointestinal disease, in particular pancreatic disease, cholecystitis, liver diseases or hepatic dysfunction.
* History of psychiatric or neurological disorders (depression, epilepsy etc.).
* Known hypersensitivity to tepotinib or its excipients.
* Presence or history of any serious allergy (requiring hospitalization or prolonged systemic treatment).
* Presence of drug or alcohol abuse, confirmed by positive test results for drugs of abuse or alcohol or history of drug and alcohol abuse in the past 3 years. Volunteers who consume more than 14 (female volunteers) or 21 (male volunteers) units of alcohol a week (unit = 1 glass of wine (125 milliliter [mL]) = 1 measure of spirits = ½ pint of beer).
* Loss or donation of more than 400 mL of blood within 12 weeks prior to entry into the trial.
* Participation in another clinical trial within the past 60 days.
* Any prescription or over the counter medication intake within 2 weeks prior to the first administration of tepotinib, including multivitamins and herbal products (St. John's wort), with the exception of acetaminophen and ibuprofen.
* Consumption of enzyme inducing or inhibiting herbal drugs, fruit juices and beverages (eg, grapefruit, grapefruit juice, Seville orange, quinine [tonic water], star fruit), and consumption of poppy seed within 3 days prior to the first administration of the investigational medicinal product.
* Excessive consumption of beverages containing xanthine (more than (>) 5 cups of coffee a day or equivalent) or inability to stop caffeine consumption while resident in the trial site. Continued use of caffeine (less than or equal to (=<)3 cups/day) or caffeine containing drinks or food, eg, coffee, tea, chocolate, Red Bull, or cola (1 caffeine unit is contained in the following items: 1 [6 ounces (oz)] cup of coffee, 2 [12 oz] cans of cola, 1 [12 oz] cup of tea, ½ [4 oz] cup of energy drink [eg, Red Bull], or 3 oz of chocolate).
* Legal incapacity or limited legal capacity.
* Unlikely to comply with the protocol requirements, instructions and trial related restrictions; eg, uncooperative attitude, inability to return for follow-up visits, and improbability of completing the trial.
* Volunteer is the Investigator or Sub-Investigator, research assistant, pharmacist, trial coordinator, other staff or relative thereof directly involved in the conduct of the trial.
* Vulnerable volunteers (eg, persons kept in detention).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2016-01-31 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2016-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Responsible, Study Director — Merck KGaA, Darmstadt, Germany
Locations (1):
- For Recruiting Locations outside US, please Contact Merck KGaA Communication Center, Darmstadt, Germany

REFERENCES:
- See also: Redacted Clinical study report, redacted clinical study protocol and redacted statistical analysis plan for this study is also available at the HC-PRCI portal (Health Canada-Public release of clinical information) — https://clinical-information.canada.ca/ci-rc/item/242300

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Overall, 65 subjects were screened for this study. Of which, 24 subjects were randomized into the study.
Groups:
- First Tepotinib Test, Then Tepotinib Reference: Subjects received a single oral dose of test treatment of film-coated tepotinib tablet (1*500 milligram [mg]) in Treatment period 1 (Day 1) followed by a single oral dose of reference treatment of film-coated tepotinib tablet (5*100 mg tablet) in Treatment period 2 (Day 22). A washout period of 21 days was maintained between the 2 treatment periods.
- First Tepotinib Reference, Then Tepotinib Test: Subjects received a single oral dose of reference treatment of film-coated tepotinib tablet (5*100 mg tablet) in Treatment period 1 (Day 1) followed by a single oral dose of test treatment of film-coated tepotinib tablet (1*500 mg) in Treatment period 2 (Day 22). A washout period of 21 days was maintained between the 2 treatment periods.
Period: Treatment Period 1 (Day 1)
Arm/Group | First Tepotinib Test, Then Tepotinib Reference | First Tepotinib Reference, Then Tepotinib Test
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Washout Period (21 Days)
Arm/Group | First Tepotinib Test, Then Tepotinib Reference | First Tepotinib Reference, Then Tepotinib Test
Started | 12 | 12
Completed | 11 | 11
Not Completed | 1 | 1
Not completed — Adverse Event | 1 | 1
Period: Treatment Period 2 (Day 22)
Arm/Group | First Tepotinib Test, Then Tepotinib Reference | First Tepotinib Reference, Then Tepotinib Test
Started | 11 | 11
Completed | 11 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The safety analysis set (SAF) included all subjects who received at least one dose of the Investigational Medicinal Product (IMP) and had follow up safety data.
Groups:
- Entire Study Population: All subjects who received a single oral dose of test treatment of film-coated tepotinib tablet (1*500 mg) or a single oral dose of reference treatment of film-coated tepotinib tablet (5*100 mg tablet) in either Treatment Period 1 or 2.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.8 (10.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 24

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to the Last Sampling Time (AUC0-t) at Concentration at or Above Lower Limit of Quantitation (LLOQ) of Tepotinib
Description: AUC0-t was calculated according to the mixed log linear trapezoidal rule.
Time Frame: Pre-dose, 0.25, 0.50, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 16, 24, 30, 36, 48, 54, 60, 72, 96, 120, 144, 168, 216, 288, 336, and 504 hours post-dose during Treatment Periods 1 and 2
Population: The pharmacokinetic (PK) analysis set included all subjects who received at least 1 dose of IMP and had at least 1 post-dose PK measurement without important protocol deviations/violations or events that could have affected the PK. Here 'Overall number of participants analyzed' = overall number of subjects evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms*hour per milliliter (ng*h/mL)
Groups:
- Tepotinib Test Treatment: Subjects who received a single oral dose of test treatment of film-coated tepotinib tablet (1*500 mg tablet) in either Treatment period 1 or 2.
- Tepotinib Reference Treatment: Subjects who received a single oral dose of reference treatment of film-coated tepotinib tablet (5*100 mg tablet) in either Treatment period 1 or 2.
Arm/Group | Tepotinib Test Treatment | Tepotinib Reference Treatment
Number analyzed (Participants) | 23 | 23
nanograms*hour per milliliter (ng*h/mL) | 25159.2 (27.0) | 25983.7 (24.0)
Statistical Analysis 1: Comparison: Tepotinib Test Treatment vs Tepotinib Reference Treatment; Test type: Superiority or Other; Geometric Least square (LS) mean ratio = 98.68, 90% CI 2-sided [93.67 to 103.96]

2. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinity (AUC0-inf) of Tepotinib
Description: AUC0-inf was calculated as AUC0-t + AUCextra. AUCextra represents the extrapolated part of AUC0-inf calculated by Clastcalc/λz, where Clastcalc was the calculated plasma concentration at the last sampling time point at which the measured plasma concentration was at or above the LLOQ and λz was the apparent terminal rate constant determined from the terminal slope of the log-transformed plasma concentration curve.
Time Frame: as for outcome 1
Population: The PK analysis set included all subjects who received at least 1 dose of IMP and had at least 1 post-dose PK measurement without important protocol deviations/violations or events that could have affected the PK. Here 'Overall number of participants analyzed' = overall number of subjects evaluable for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Tepotinib Test Treatment | Tepotinib Reference Treatment
Number analyzed (Participants) | 18 | 17
ng*h/mL | 25709.6 (29.6) | 26990.3 (26.1)
Statistical Analysis 1: Comparison: Tepotinib Test Treatment vs Tepotinib Reference Treatment; Test type: Superiority or Other; Geometric LS mean ratio = 95.71, 90% CI 2-sided [88.43 to 103.59]

3. Primary Outcome: Maximum Plasma Concentration Observed (Cmax) of Tepotinib
Description: Cmax was obtained directly from the concentration versus time curve.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Tepotinib Test Treatment | Tepotinib Reference Treatment
Number analyzed (Participants) | 23 | 23
ng/mL | 463.0 (26.2) | 486.3 (19.8)
Statistical Analysis 1: Comparison: Tepotinib Test Treatment vs Tepotinib Reference Treatment; Test type: Superiority or Other; Geometric LS mean ratio = 96.88, 90% CI 2-sided [90.8 to 103.36]

4. Primary Outcome: Time to Reach the Maximum Plasma Concentration (Tmax) of Tepotinib
Description: Time to reach the maximum plasma concentration (Tmax) was obtained directly from the concentration versus time curve.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Tepotinib Test Treatment | Tepotinib Reference Treatment
Number analyzed (Participants) | 23 | 23
hours | 8.000 [4.00 to 24.00] | 8.000 [4.00 to 16.00]
Statistical Analysis 1: Comparison: Tepotinib Test Treatment vs Tepotinib Reference Treatment; Test type: Superiority or Other; p = 0.8981, Wilcoxon signed-rank test; Median Difference (Net) = 0.000, 90% CI 2-sided [-1.000 to 1.025]

5. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to the Last Sampling Time (AUC0-t) of Tepotinib Metabolites (MSC2571109A and MSC2571107A)
Description: AUC0-t at which the concentration was at or above LLOQ was calculated according to the mixed log linear trapezoidal rule.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Tepotinib Test Treatment | Tepotinib Reference Treatment
Number analyzed (Participants) | 23 | 23
ng*h/mL
  MSC2571109A | 13637.3 (30.4) | 14164.7 (27.1)
  MSC2571107A | 846.2 (42.4) | 849.5 (36.3)

6. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinity (AUC0-inf) of Tepotinib Metabolites (MSC2571109A and MSC2571107A)
Description: as for outcome 2
Time Frame: as for outcome 1
Population: The PK analysis set. Here 'Overall number of participants analyzed' = overall number of subjects evaluable for this outcome measure and "Number Analyzed" signifies those subjects who were evaluable for specified category.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Tepotinib Test Treatment | Tepotinib Reference Treatment
Number analyzed (Participants) | 21 | 22
ng*h/mL
  MSC2571109A | 13932.6 (31.0) | 14541.7 (25.5)
  MSC2571107A: number analyzed (Participants) | 20 | 20
  MSC2571107A | 865.0 (39.7) | 830.4 (35.6)

7. Secondary Outcome: Maximum Plasma Concentration Observed (Cmax) of Tepotinib Metabolites (MSC2571109A and MSC2571107A)
Description: Cmax was obtained directly from the concentration versus time curve.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Tepotinib Test Treatment | Tepotinib Reference Treatment
Number analyzed (Participants) | 23 | 23
ng/mL
  MSC2571109A | 160.40 (28.6) | 160.86 (24.4)
  MSC2571107A | 11.630 (38.2) | 11.299 (29.9)

8. Secondary Outcome: Time to Reach the Maximum Plasma Concentration (Tmax) of Tepotinib Metabolites (MSC2571109A and MSC2571107A)
Description: Tmax was obtained directly from the concentration versus time curve.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Tepotinib Test Treatment | Tepotinib Reference Treatment
Number analyzed (Participants) | 23 | 23
hours
  MSC2571109A | 24.00 [24.0 to 48.0] | 24.02 [24.0 to 97.3]
  MSC2571107A | 24.00 [16.0 to 48.0] | 24.00 [16.0 to 48.0]

9. Secondary Outcome: Apparent Terminal Half-Life (t1/2) of Tepotinib and Metabolites (MSC2571109A and MSC2571107A) in Plasma
Description: t1/2 was defined as the time taken for the plasma concentration or the amount of drug in the body to be reduced by half.
Time Frame: as for outcome 1
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Tepotinib Test Treatment | Tepotinib Reference Treatment
Number analyzed (Participants) | 21 | 22
hours
  Tepotinib: number analyzed (Participants) | 18 | 17
  Tepotinib | 35.27 (18.1) | 34.27 (22.5)
  MSC2571109A | 47.33 (25.4) | 46.39 (28.8)
  MSC2571107A: number analyzed (Participants) | 20 | 20
  MSC2571107A | 42.39 (17.0) | 40.18 (21.3)

10. Secondary Outcome: Apparent Terminal Rate Constant (λz) of Tepotinib and Metabolites (MSC2571109A and MSC2571107A) in Plasma
Description: Apparent terminal rate constant was determined from the terminal slope of the log-transformed plasma concentration curve using linear regression on terminal data points of the curve.
Time Frame: as for outcome 1
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: 1/h
Arm/Group | Tepotinib Test Treatment | Tepotinib Reference Treatment
Number analyzed (Participants) | 21 | 22
1/h
  Tepotinib: number analyzed (Participants) | 18 | 17
  Tepotinib | 0.019652 (18.1) | 0.020229 (22.5)
  MSC2571109A | 0.014643 (25.4) | 0.014942 (28.8)
  MSC2571107A: number analyzed (Participants) | 20 | 20
  MSC2571107A | 0.016350 (17.0) | 0.017252 (21.3)

11. Secondary Outcome: Total Body Clearance of Drug From Plasma (CL/f) for Tepotinib
Description: CL/f following oral administration was calculated as Dose/AUC0-inf, where AUC0-inf calculated as AUC0-t + AUCextra. AUCextra represents the extrapolated part of AUC0-inf calculated by Clastcalc/λz, where Clastcalc was the calculated plasma concentration at the last sampling time point at which the measured plasma concentration was at or above the LLOQ and λz was the apparent terminal rate constant determined from the terminal slope of the log-transformed plasma concentration curve.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liter/hour
Arm/Group | Tepotinib Test Treatment | Tepotinib Reference Treatment
Number analyzed (Participants) | 18 | 17
liter/hour | 17.503 (29.6) | 16.673 (26.1)

12. Secondary Outcome: Apparent Volume of Distribution (Vz/f) for Tepotinib
Description: Vz/f is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Vz/f during the terminal phase was reported.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: liters
Arm/Group | Tepotinib Test Treatment | Tepotinib Reference Treatment
Number analyzed (Participants) | 18 | 17
liters | 890.7 (27.7) | 824.2 (21.4)

13. Secondary Outcome: Extrapolated Area Under the Plasma Concentration-Time Curve From Time t to Infinity (%AUCextra) of Tepotinib and Metabolites (MSC2571109A and MSC2571107A)
Description: %AUCextra was defined as a percentage of AUC0-inf obtained by extrapolation: %AUCextra = (1- [AUC0-t / AUC0-inf])*100. %AUCextra was reported in terms of percentage of AUC0-inf.
Time Frame: as for outcome 1
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of AUC0-inf
Arm/Group | Tepotinib Test Treatment | Tepotinib Reference Treatment
Number analyzed (Participants) | 21 | 22
percentage of AUC0-inf
  Tepotinib: number analyzed (Participants) | 18 | 17
  Tepotinib | 1.5025 (36.7) | 1.5394 (44.7)
  MSC2571109A | 0.4040 (45.9) | 0.4257 (48.1)
  MSC2571107A: number analyzed (Participants) | 20 | 20
  MSC2571107A | 0.9715 (49.1) | 0.9748 (46.3)

14. Secondary Outcome: Ratio of Area Under the Plasma Concentration-Time Curve From Time Zero to Infinity (AUC0-inf) of Metabolite (MSC2571109A or MSC2571107A) to AUC0-inf of Tepotinib
Description: Ratio of AUC0-inf of Metabolite (MSC2571109A or MSC2571107A) to AUC0-inf of tepotinib was reported.
Time Frame: as for outcome 1
Population: as for outcome 6
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Tepotinib Test Treatment | Tepotinib Reference Treatment
Number analyzed (Participants) | 21 | 22
ratio
  MSC2571109A | 0.5362 (16.3) | 0.5353 (18.0)
  MSC2571107A: number analyzed (Participants) | 20 | 20
  MSC2571107A | 0.03397 (25.9) | 0.03216 (22.0)

15. Secondary Outcome: Ratio of Maximum Plasma Concentration Observed (Cmax) of Metabolite (MSC2571109A or MSC2571107A) to Cmax of Tepotinib
Description: Ratio of Cmax of metabolite (MSC2571109A or MSC2571107A) to Cmax of tepotinib was reported.
Time Frame: as for outcome 1
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Tepotinib Test Treatment | Tepotinib Reference Treatment
Number analyzed (Participants) | 23 | 23
ratio
  MSC2571109A | 0.3464 (22.4) | 0.3308 (23.4)
  MSC2571107A | 0.02512 (29.0) | 0.02323 (29.3)

16. Secondary Outcome: Number of Subjects With Treatment-emergent Adverse Events (TEAEs), Serious TEAEs, TEAEs Leading to Death, TEAEs Leading to Discontinuation
Description: An adverse event (AE) was defined as any untoward medical occurrence in a subject which does not necessarily have a causal relationship with the treatment. An AE was any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with use of a medicinal product, whether or not considered related to the medicinal product. A serious adverse event (SAE) was an AE that resulted in any of the following outcomes: death; life threatening; persistent/significant disability/incapacity; initial or prolonged inpatient hospitalization; congenital anomaly/birth defect or was otherwise considered medically important. The term TEAE is defined as AEs starting or worsening after the first intake of the study drug.
Time Frame: Baseline up to end of trial (up to Day 43)
Population: SAF population. A total of 24 subjects were evaluated for adverse events. Because 1 subject in each treatment sequence discontinued before receiving the second treatment, only 23 subjects received Test Treatment and 23 subjects received Reference Treatment.Thus, number of subjects analyzed per treatment is mentioned as 23.
Measure: Count of Participants; unit: Participants
Arm/Group | Tepotinib Test Treatment | Tepotinib Reference Treatment
Number analyzed (Participants) | 23 | 23
Participants
  TEAEs | 10 | 9
  Serious TEAEs | 0 | 0
  TEAEs Leading to Death | 0 | 0
  TEAE leading to Discontinuation | 1 | 1

17. Secondary Outcome: Number of Subjects With Clinically Significant Change From Baseline in Vital Signs, Electrocardiogram (ECG) and Laboratory Parameters
Description: Number of subjects with clinically significant change from baseline in vital signs, ECG and laboratory parameters were reported. Clinical Significance was decided by the investigator. Vital signs included oral body temperature, systolic blood pressure, diastolic blood pressure, and pulse rate. The 12-lead ECGs were recorded after the subjects have rested for at least 5 minutes in supine position. The parameters included heart rate (HR), RR, PR, QRS, QT and QTcB calculated by the Bazett formula. Laboratory investigation included hematology, biochemistry, urinalysis, and coagulation.
Time Frame: Baseline up to end of trial (up to Day 43)
Population: SAF population. A total of 24 subjects were evaluated for adverse events. Because 1 subject in each treatment sequence discontinued before receiving the second treatment, only 23 subjects received Test Treatment and 23 subjects received Reference Treatment. Thus, number of subjects analyzed per treatment is mentioned as 23.
Measure: Count of Participants; unit: Participants
Arm/Group | Tepotinib Test Treatment | Tepotinib Reference Treatment
Number analyzed (Participants) | 23 | 23
Participants
  Vital Signs | 0 | 0
  ECG Values | 0 | 0
  Laboratory Values | 0 | 0

ADVERSE EVENTS:
Time Frame: Baseline up to end of trial (up to Day 43)
Description: The safety analysis set included all subjects who received at least 1 dose of the IMP and had follow up safety data. A total of 24 subjects were evaluated for adverse events. Because 1 subject in each treatment sequence discontinued before receiving the second treatment, only 23 subjects received Test Treatment and 23 subjects received Reference Treatment. Thus, number of subjects analyzed per treatment is mentioned as 23.
Arm/Group | Tepotinib Test Treatment | Tepotinib Reference Treatment
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 10/23 | 9/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tepotinib Test Treatment (N=23) | Tepotinib Reference Treatment (N=23)
Arthropod Bite (Injury, poisoning and procedural complications) | 1 | 0
Foreign Body In Eye (Injury, poisoning and procedural complications) | 0 | 1
Amylase Increased (Investigations) | 1 | 0
Lipase Increased (Investigations) | 1 | 0
Dry Throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0
Catheter Site Inflammation (General disorders) | 1 | 0
Catheter Site Related Reaction (General disorders) | 0 | 2
Chills (General disorders) | 0 | 1
Influenza Like Illness (General disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Dyspepsia (Gastrointestinal disorders) | 1 | 0
Mouth Ulceration (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Toothache (Gastrointestinal disorders) | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 1
Hepatic Function Abnormal (Hepatobiliary disorders) | 1 | 0
Dermatitis Contact (Skin and subcutaneous tissue disorders) | 2 | 0
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 1
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 0 | 2
Influenza (Infections and infestations) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publications and presentations of the results (abstracts in journals or newspapers, oral presentations, etc.), either in whole or in part, by Investigators or their representatives will require review by the Sponsor before submission. The Sponsor will not suppress publication, but maintains the right to delay publication in order to protect intellectual property rights.